CLINICAL TRIAL: NCT04467801
Title: A Multi-center Phase II Study of Ipatasertib in Combination With Docetaxel in Metastatic/Advanced NSCLC Patients Who Have Failed or Are Intolerant to 1st Line Immunotherapy (Ipat-Lung)
Brief Title: Ipatasertib and Docetaxel in Metastatic NSCLC Patients Who Have Failed 1st Line Immunotherapy
Acronym: Ipat-Lung
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jun Zhang, MD, PhD (Other)
Collaborators: University of Iowa (Other); University of Kentucky (Other)
Responsible Party: Sponsor-Investigator, Jun Zhang, MD, PhD, MD, PhD, University of Kansas Medical Center
Organization: University of Kansas Medical Center (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IIT-2019-IpatTax
Record Dates: First submitted 2020-06-15; First posted 2020-07-13 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-11

CONDITIONS: NSCLC Stage IV; NSCLC Stage IIIB
Keywords: Advanced/metastatic NSCLC
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — ipatasertib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (Experimental): Ipatasertib, 400 mg once daily, Oral, Days 1-14 of each 21 day cycle (2 weeks on and 1 week off).
  Docetaxel, 75 mg/m2, Intra-venous, Day 1 of each 21 day cycle.
  Interventions: Drug: Ipatasertib

INTERVENTIONS:
Drug: Ipatasertib — Ipatasertib is a novel ATP-competitive inhibitor. It is taken by mouth once daily.

SUMMARY:
For metastatic/advanced NSCLC patients who do not have targetable mutations, either immunotherapy targeting the programmed death-1 and its ligand (PD-1/L1) pathway alone or in combination with platinum doublet chemotherapy is now a standard of care. However, still about half of the patients do not benefit due to treatment resistance. It is therefore critically important to find novel therapies and combinations to benefit patients who have failed or are intolerant to 1st line immunotherapy.

This study hypothesizes that ipatasertib in combination with taxane (e.g. docetaxel) can be an effective strategy. Ipatasertib is a novel adenosine triphosphate (ATP)-competitive inhibitor that has demonstrated robust and selective targeting of protein kinase B (PKB, also known as AKT) in cancer patients. Importantly, evidence from preclinical studies has demonstrated that AKT inhibitors (e.g. ipatasertib) can enhance the therapeutic effect of chemotherapy as well as immunotherapy via modulating Phosphatidylinositol 3-kinase (PI3'K)-AKT activity.

ELIGIBILITY:
Inclusion Criteria:

* Ability of participant OR Legally Authorized Representative (LAR) to understand this study, and participant or LAR willingness to sign a written informed consent
* Life expectancy ≥12 weeks
* Males and females age ≥ 18 years
* Allowable type and amount of prior therapy:

First line anti-Programmed death receptor and ligand (PD1/PD-L1), either single agent or in combination with chemotherapy

* Eastern Cooperative Oncology Group (ECOG) Performance Status 0 or 1
* Measurable disease per RECIST version 1.1
* Diagnoses of advanced/metastatic NSCLC and have failed or are intolerant to 1st line anti-PD1/PD-L1, either single agent or in combination with chemotherapy, and have either exhausted or decline or not be candidates for all available standard of care therapies.
* Adequate organ function
* Women of child-bearing potential and men with partners of child-bearing potential must agree to practice sexual abstinence, or to use an acceptable form of contraception for the duration of study participation, and for 90 days following completion of therapy
* Men of child-bearing potential must agree not to donate sperm while on this study and for 90 days after their last study treatment

Exclusion Criteria:

* Is not concurrent enrolled in another clinical study, unless it is an observational (non-interventional) clinical study or if the participant is in the follow-up period of an interventional study
* Is not currently on or is not anticipated to use other investigational agents within 14 days prior to and while participating in this study
* Does not have mixed small cell and non-small cell lung cancer histology
* Does not have any unresolved toxicity CTCAE >Grade 2 from the prior 1st immunotherapy. Patients with irreversible toxicity that is not reasonably expected to be exacerbated by study drug may be included
* Patients who have targetable mutations that qualify for targeted therapy (e.g. mutations of epidermal growth factor receptor (EGFR), serine/ threonine- protein kinase (BRAF), anaplastic lymphoma kinase (ALK), tyrosine- protein kinase (ROS1), neurotrophic receptor tyrosine kinase (NTRAK)) will be excluded from this study
* Is not on concomitant therapy intended for the treatment of cancer (including, but not limited to, chemotherapy, hormonal therapy, immunotherapy, radiotherapy, and herbal therapy) for 14 days prior to starting study treatment, depending on the agent and during study treatment, until disease progression is documented and the patient has discontinued study treatment, with the exception of palliative radiotherapy and local therapy per PI discretion
* Does not chronically use a strong cytochrome P4503A4 (CYP3A4/5) inhibitor or inducer, or sensitive CYP3A substrates with a narrow therapeutic window
* Has not had recent major surgery within 4 weeks prior to entry into the study (excluding the placement of vascular access) that would prevent administration of study drug
* Does not have uncontrolled systemic disease
* Does not have uncontrolled brain metastasis
* Does not have history of allergy to taxanes
* Does not have history of leptomeningeal carcinomatosis
* Does not have recent history of myocardial infarction (MI) or symptomatic coronary artery disease within 6 months of screening
* Is not receiving active therapy for HIV, hepatitis B or hepatitis C
* Does not have history of malabsorption syndrome or other condition that would interfere with enteral absorption or results in the inability or unwillingness to swallow pills
* Does not have history of Type I or Type II diabetes mellitus requiring insulin (Patients who are on a stable dose of oral diabetes medication greater than or equal to 2 weeks prior to initiation of study treatment
* Does not have Grade greater than or equal to 2 uncontrolled or untreated hypercholesterolemia or hypertriglyceridemia
* Does not have history of or active inflammatory bowel disease (e.g., Crohn's disease and ulcerative colitis) or active bowel inflammation (e.g., diverticulitis)
* Does not have active pneumonitis
* Does not have history of lung disease: interstitial lung disease, idiopathic pulmonary fibrosis, cystic fibrosis, Aspergillosis, active tuberculosis, or history of opportunistic infections
* Does not have uncontrolled pleural effusion/pericardial effusion/or ascites as determined by the investigator
* Does not have active ventricular arrhythmia requiring medication
* Does not have psychiatric illness/social situations that would limit compliance with study requirements or compromise the ability of the patient to give written informed consent
* Is not pregnant, breast feeding or planning to become pregnant while receiving study treatment or for less than 90 days after the last dose of study treatment
* For males with partners of childbearing potential, is not planning to father a child or donate sperm while receiving study treatment or for less than 90 days after the last dose of study treatment
* Does not have any condition that, in the opinion of the investigator, would interfere with evaluation or interpretation of patient safety or study results

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2021-09-14 (Actual); Primary Completion 2024-08 (Estimated); Study Completion 2025-08 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | up to 12 months
  RECIST 1.1

SECONDARY OUTCOMES:
Number of adverse events experienced by participants receiving treatment with ipatasertib in combination with docetaxel | At cycle 1day 8 (each cycle is 21 days) up to 2 months (60 days) after End of treatment
  CTCAE Version 5.0
Overall Response Rate | every 6 weeks up to 12 months
  RECIST 1.1
Overall Survival | Cycle 1day 1 (each cycle is 21 days) to up to 12 months after end of treatment
  Medical record

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, PhD, Principal Investigator — The University of Kansas
Locations (5):
- United States (5):
  - The University of Kansas Cancer Center (KUCC), Fairway, Kansas
  - The University of Kansas Cancer Center, Westwood Campus, Kansas City, Kansas
  - The University of Kansas Cancer Center, Overland Park Clinic, Overland Park, Kansas
  - The University of Kansas Cancer Center, North Clinic, Kansas City, Missouri
  - The University of Kansas Cancer Center, Lee's Summit Clinic, Lee's Summit, Missouri

IPD SHARING:
Plan to Share IPD: No